CLINICAL TRIAL: NCT04916717
Title: Effect Of Counselıng on Qualıty of Lıfe and Self-Care Agency for Patıents Who Are Scheduled for Total Knee Replacement
Brief Title: Effect Of Counselıng
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uşak University (Other)
Responsible Party: Principal Investigator, çiğdem kaya, Lecturer, PhD, Uşak University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: ckaya
Record Dates: First submitted 2021-05-27; First posted 2021-06-07 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Total Knee Replacement; Quality of Life; Nursing Caries
Keywords: total knee replacement; nursing counseling; counseling; quality of life; self care agency
MeSH Terms: interventions — Counseling; Patient Education as Topic

STUDY DESIGN:
Intervention Model Description: This is a quantitative study and has a quasi-experimental design with a control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Counseling (Other): Quasi-experimental design. Face-to-face and telephone counseling were applied to individuals in the intervention group.
  Interventions: Other: Counseling

INTERVENTIONS:
Other: Counseling — Face-to-face and telephone counseling were applied to individuals in the intervention group.
  Other Names: Patient education

SUMMARY:
This study aims to determine the effect of counseling on quality of life and self-care agency for patients who are scheduled for TKR.

DETAILED DESCRIPTION:
This is a quantitative study and has a quasi-experimental design with a control group. The sample of the study consisted of 79 patients including intervention (n=39) and control (n=40). The data are collected by the face-to-face interview method using Patient Identification Form, Quality of Life Scale, and Self-Care Agency Scale before surgery, and 6-8th weeks after discharge. Face-to-face and telephone counseling were applied to individuals in the intervention group. The x2, t-test, one-factor variance analysis, and two-factor variance analysis were used in the analysis of the data.

ELIGIBILITY:
Inclusion Criteria:

* undergoing TKA for the first time, being scheduled to have unilateral TKA, having surgery for osteoarthritis, having no postoperative complications, fulfilment of discharge criteria after surgery, being aged 18 years or older, being conscious, orientation to place and time, having no hearing or speech problems, ability to understand and speak Turkish, being at least literate, not being diagnosed with any psychiatric diseases and not having a history of cancer.

Exclusion Criteria:

* diagnoses of neurological (e.g. Alzheimer's disease) and psychiatric disorders (e.g. schizophrenia) likely to affect cognitive functions, first accepting to participate in the study and then dropping out of the study, development of complications during follow-up (e.g. infection), unavailability when called and lost to follow-up.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Quality of life (SF-36) | up to 16 weeks
  in quality of life change from the preoperative period to 6-8th weeks and 14-16th weeks (postoerative period)
Self Care Agency | up to16 weeks
  in self care agency change from the preoperative period to 6-8th weeks and 14-16th weeks (postoerative period)

CONTACTS AND LOCATIONS:
Locations (1):
- Usak University Education and Research Hospital, Uşak, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided